CLINICAL TRIAL: NCT00850798
Title: The Benefits of Intensive Glycemic Control in Elderly Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Chen-Hsen Lee, Chairman, Institutional Review Board, Taipei Veterans General Hospital,Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHIRB 97-12-04
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Elder patients; Glycemic control; Men or women aged ≥80 years at time of randomization. There is no upper age limit.; Be able to walk by themselves; They had their first diagnosis of type 2 diabetes mellitus at age 30 years or older.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fasting plasma glucose (mg/dL) 90 to 130 Glycated hemoglobin (%) 6.0 to 7.0
  Interventions: Drug: Intensive glycemic control
- 2 (Active Comparator): Fasting plasma glucose (mg/dL) 90 to 180 Glycated hemoglobin (%) 7.0 to 9.0
  Interventions: Drug: Conservative glycemic control

INTERVENTIONS:
Drug: Intensive glycemic control — Intensive glycemic control
  Arms: 1
Drug: Conservative glycemic control — OADs and insulin
  Arms: 2

SUMMARY:
Aims/hypothesis:

Populations worldwide are aging and type 2 diabetes is common in individuals aged >80 years. The important issue that needs to be considered is whether tight glycemic control is benefits for elderly patients with type 2 diabetes. The benefits of intensive glucose control remain uncertain for the heterogeneous population of older diabetic patients due to a lack of clinical trial data evaluating the benefits of long-term intensive glucose control in older patients. This study is designed to provide reliable evidence on the balance of benefits and risks conferred by intensive glucose control in elderly patients with type 2 diabetes Methods: This is a prospective, randomized, open-labeled, controlled design to assess the benefits of treating elderly patients with type 2 diabetes. The study will include 208 elderly patients with type 2 diabetes and follow-up for 5 years. Eligible patients are randomized to receive intensive (A1C <7.0%) or conservative (A1C around 8.0%) glycemic control. The primary study outcomes are a composite of macrovascular events and a composite of microvascular events, considered both jointly and separately. The secondary outcomes are death from any cause, death from cardiovascular causes, total coronary events, total cerebrovascular events, heart failure, peripheral vascular events, all cardiovascular events, and hospitalization for 24 hours or more.

Expected results: This study is designed to provide reliable evidence on the balance of benefits and risks conferred by intensive and conservative glucose control in elderly patients with type 2 diabetes. Once completed, this trial will clearly influence the management of elderly patients with type 2 diabetes, regardless of the results.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥80 years at time of randomization.There is no upper age limit.
* Be able to walk by themselves
* They had their first diagnosis of type 2 diabetes mellitus at age 30 years or older.

Exclusion Criteria:

* Known advanced diabetic complications (such as proliferative retinopathy, chronic kidney disease stage IV or above).
* Overt clinical congestive heart failure (CHF) requiring treatment with a diuretic or ACE inhibitor.
* Previous documented cerebral or subarachnoid haemorrhage in the last 6 months
* Condition expected to severely limit survival
* Clinical diagnosis of dementia
* Resident in a nursing home

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The primary study outcomes are a composite of macrovascular events and a composite of microvascular events, considered both jointly and separately. | Every 6 months and up to 5 years

SECONDARY OUTCOMES:
The secondary outcomes are death from any cause, disability from any cause, total coronary events, total cerebrovascular events, heart failure, peripheral vascular events, all cardiovascular events, and hospitalization for 24 hours or more. | Every 6 months and upto 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chen-Hsen Lee, Taipei, Taiwan